CLINICAL TRIAL: NCT01938053
Title: Improving Sexually Transmitted Infection (STI) Results Notification and Partner Services
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: University of Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: K12HD051953 Reed; K12HD051953 (NIH)
Record Dates: First submitted 2013-09-05; First posted 2013-09-10 (Estimated); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Sexually Transmitted Infections
Keywords: STI, STD
MeSH Terms: conditions — Sexually Transmitted Diseases | interventions — CD56 Antigen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Reminder card with no number (Other): Patients receive a card to remind them of the time frame for results but no number is listed.
  Interventions: Other: Call when test results are ready; Other: Text message when test results are ready; Other: Call and text message when test results are ready
- Card with number (Other): Patients receive a card to remind them of the time frame for results but and a number to call for results is listed
  Interventions: Other: Call when test results are ready; Other: Text message when test results are ready; Other: Call and text message when test results are ready

INTERVENTIONS:
Other: Call when test results are ready — Patients are called when the test results are ready
Other: Text message when test results are ready — Patients receive a text message when results are ready
Other: Call and text message when test results are ready — Patients receive both a call and a text message when test results are resay

SUMMARY:
The primary goal of this project is to improve the process for contacting patients that test positive for a sexually transmitted infection (STI) in the emergency department by using text messaging. We believe patients that are contacted by both a phone call and a text message will be reached more often and they will be reached sooner than those that only receive a phone call or only a text message. In addition, patients will be given reminder cards at the time of testing to remind them that they will be contacted within 7 days if they test positive. Half of the reminder cards will have a number to call for test results. We believe patients that receive a card with a number are more likely to be contacted within 7 days.

DETAILED DESCRIPTION:
Aim 1: To improve the results notification system among all female adolescents who test positive for STIs in the ED using mobile phone texting technology.

Hypothesis 1: We will increase our contact rate for STI positive adolescents in the ED from 65-82%.

Hypothesis 2: We will decrease the time interval between testing and appropriate STI treatment by the ED.

Hypothesis 3: We will decrease the recidivism rates for STI positive patients diagnosed in the ED.

Aim 2: To explore qualitatively the barriers to and preferences for partner notification and treatment among 14-21 year-old females and males being tested for STIs in the ED.

Aim 3: To determine baseline rates of partner notification and preferences around partner notification among STI-positive females in the ED, and to explore the feasibility of ED personnel notifying their sexual partners.

ELIGIBILITY:
Inclusion Criteria:

* 14 to 21 years old
* Seen in the emergency department at Cincinnati Children's Hospital Medical Center
* Test positive for an STI

Exclusion Criteria:

* Seen for a psychiatric evaluation
* Seen for sexual assault or abuse

Ages: 14 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 609 (Actual)
Dates: Start 2011-04; Primary Completion 2013-06 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Contact rate | 7 days
  The percentage of patients that are contacted within 7 days of their emergency department visit

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Reed, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States